CLINICAL TRIAL: NCT04827511
Title: Refractive Disorders and Seric Vitamin D Level in Children With Disabilities
Acronym: REDIC
Status: Completed | Type: Observational
Sponsor: Holhos Larisa Bianca (Other)
Responsible Party: Sponsor-Investigator, Holhos Larisa Bianca, Specialist in Ophthalmology, Elisantes Teola SRL
Organization: Elisantes Teola SRL (Other)
Other Study IDs: 142312202069
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Child, Only
Keywords: disability, healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 19 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cohort group: 80 children with disabilities like autism, ADHD, Down syndrome, deafness, phocomelia, dyslexia, different motor problems
  Interventions: Other: Refraction measurement with auto-ref-keratometer Canon
- control group: 81 healthy children, not known or diagnosed with a chronic disease of any kind
  Interventions: Other: Refraction measurement with auto-ref-keratometer Canon

INTERVENTIONS:
Other: Refraction measurement with auto-ref-keratometer Canon — Refractive measurement and vitamin D level dosing

SUMMARY:
The investigator want to determine the refractive status of 80 children with disabilities and of 81 healthy children from a witness group. The vitamin D level of the children will be dosed for making different correlations with visual acuity status.

DETAILED DESCRIPTION:
Refraction measurement will be done by the investigator in all 161 children. Visual acuity is checked, initial and after correction with proper correction. Vitamin D level is dosed from all the children in order to make correlations with the visual acuity, refractive status and risk for visual impairment.

ELIGIBILITY:
Inclusion Criteria:

* children with disabilities and healthy children

Exclusion Criteria:

* children diagnosed with another chronic diseases

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 80 children with disabilities like ADHD, autism, Down syndrome, deafness, phocomelia and 81 clinically healthy children
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Refractive disorders in children with disabilities | 1 January 2019-31 August 2020
  Prevalence of refractive disorders in children with disabilities

CONTACTS AND LOCATIONS:
Overall Officials: Holhoș L Bianca, Doctor, Principal Investigator — Faculty of Medicine and Pharmacy Oradea
Locations (1):
- Holhoș Larisa Bianca, Marghita, Bihor County, Romania

IPD SHARING:
Plan to Share IPD: Yes
Reports from the statistical analysis
Supporting Information: CSR
Time Frame: 20/10/2021-20/10/2031
Access Criteria: by invitation